CLINICAL TRIAL: NCT04744220
Title: Evaluation of the Effect of Yoga Training on Functional Capacity and Quality of Life in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, salih tan, doctorate, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.19408
Record Dates: First submitted 2021-01-21; First posted 2021-02-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bronchiectasis Adult
Keywords: Yoga Training; Quality of Life; Functional Capacity; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: The cases will be randomly divided into two groups as 24 control groups and 24 yoga training groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Training Group (Experimental): Training: Before the yoga program, the patients will be informed about the bronchiectasis disease and its symptoms, as well as all the parameters used in the evaluation, tests and the content of the yoga session.
  During the program, the perceived fatigue intensity of the patients will be questioned with the Modified Borg Scale.
  Yoga Session
  1-8 weeks and duration
  * Breathing Exercises 5 min
  * Instant Relaxation Technique 2 min
  * Warm-up Exercises 10 min
  * Quick Relaxation Technique 3 min
  * Asanas (Posture Exercises) 15 min
  * Alternative Breathing Exercises 10 min
  * Deep Relaxation Technique 3 min
  Interventions: Other: Yoga Training Program (exercises)
- Control group (No Intervention): Training: The exercise program will include respiration exercises that they can do at home.
  Before the exercise program, the patients will be informed about the bronchiectasis disease and its symptoms, as well as all the parameters and tests used in the evaluation. Respiratory control, breathing exercises, relaxation techniques and the reasons, importance and effects of exercise training in the treatment program will be explained.
  Breathing Exercises (10 min) Pursed-lip breathing training, Chest breathing exercise (10 repetitions), Diaphragmatic breathing exercise (10 repetitions), Bilateral basal expansion breathing exercises (10 repetitions)

INTERVENTIONS:
Other: Yoga Training Program (exercises) — Training: Before the yoga program, the patients will be informed about the bronchiectasis disease and its symptoms, as well as all the parameters used in the evaluation, tests and the content of the yoga session. The patients will start with breathing exercises, then relaxation exercises, warm-up exercises, asanas (posture exercises) and finally the yoga training program will be completed with deep relaxation technique.
  Arms: Yoga Training Group

SUMMARY:
Evaluation of the Effect of Yoga Training on Functional Capacity and Quality of Life in Patients with Bronchiectasis between the ages of 30-55

DETAILED DESCRIPTION:
Investigating the effect of yoga training on functional capacity and quality of life and comparing with previous studies

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bronchiectasis
* Age 30-55
* Not having a known systemic, orthopedic or neurological disease

Exclusion Criteria:

* Severe heart failure
* People who had an acute exacerbation up to three weeks ago will not be included in the study

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Patient Follow-up Form | Baseline
  The demographic characteristics, physical characteristics such as age, height and body weight of the individuals included in the study and their education status will be recorded.

SECONDARY OUTCOMES:
Dyspnea Assessment | Before and after treatment (8 week)
  Dyspnea will be assessed by the modified Medical Research Council (MMRC) dyspnea scale. Individuals will be asked to choose the statement that best describes their dyspnea level.
  Scoring in MMRC varies between 0-4 points. "0 points" means that there is no dyspnea; "4 points" indicates a perception of dyspnea during basic daily life activities such as dressing.

OTHER OUTCOMES:
Respiratory Function Test | Before and after treatment( 8 week )
  A spirometer will be used to evaluate the lung function of individuals. It will be expressed as a percentage of the expected values by age, height, body weight and gender.
Quality of Life Assessment | Before and after treatment (8 week)
  Quality of life, St. George's Respiratory Questionnaire (SGRQ). SGRQ is a health-related quality of life questionnaire that questions a total of 50 items under 3 main components: symptoms (8 items), activity (16 items) and effects of disease (26 items). The symptoms component includes the frequency and duration of symptoms such as cough, sputum, shortness of breath, wheezing.
  The activity component relates to physical activities that are restricted due to shortness of breath. It includes factors such as the effects component of the disease, the drugs used and its side effects, the individual's expectations for health and the discomfort they face in daily life. The total score is between 0-100. The higher the score, the lower the quality of life
Evaluation of Functional Capacity | Before and after treatment (8 week)
  Individuals' functional capacity will be evaluated with the six-minute walking test (6MWT). During the 6MWT, individuals are asked to walk in a straight corridor of 30 meters as fast as possible, at their own walking pace in standard directions.
  At the end of the test, the walking distance is recorded in meters.
Assessment of Sleep Quality | Before and after treatment (8 week)
  Pittsburgh Sleep Quality Index (PSQI) will be used to evaluate the sleep quality of the individuals participating in our study before and after the 8-week study period.
  PSQI is a test that plays a role in determining sleep quality and sleep-related disorders in the last month. It is a scale consisting of 19 self-report items, a total of 24 questions with a score range of 0-21, and the remaining five questions must be answered by a roommate or a spouse. It is a test that evaluates a wide variety of areas related to sleep quality, including components, sleep time, delays in falling asleep, the frequency and severity of sleep-related problems, and the impact of poor sleep on an individual's work.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Tan, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No